CLINICAL TRIAL: NCT03492632
Title: Ovarian Reserve in Patients With Psoriasis
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berna Aslan Cetin, Principle investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2017/325
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Psoriasis; Anti Mullerian Hormone; Ovarian Reserve
Keywords: psoriasis; Anti mullerian hormone; ovarian reserve; antral follicle count
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for the measurement of serum FSH,LH,E2,PRL and AMH
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with Psoriasis: Reproductive age women newly diagnosed with psoriasis
  Interventions: Other: Hormone panel
- Women without Psoriasis: Reproductive age women without psoriasis to serve as control
  Interventions: Other: Hormone panel

INTERVENTIONS:
Other: Hormone panel — Blood sampling on the 3rd day of menstrual cycle for the measurement of serum FSH,LH,PRL,E2 and AMH hormone levels.

SUMMARY:
Psoriasis is a common autoimmune disease. It affects women of all ages including reproductive years. Autoimmune diseases including psoriasis are linked to premature ovarian reserve. This study aims to measure serum hormones including FSH,LH,E2,PRL and AMH (indicators of ovarian reserve) in women with and without psoriasis.

DETAILED DESCRIPTION:
Psoriasis is a common autoimmune disease. It affects women of all ages including reproductive years. Almost 75% of patients are diagnosed before the age of 40. There is also increased evidence on autoimmune disease and their link to premature ovarian failure.Ovarian reserve is important for the reproductive period. The measurements of serum hormones including follicle stimulating hormone (FSH),luteinizing hormone (LH),prolactin (PRL), estradiol (E2) and anti-mullerian hormone (AMH) will give us an idea about the ovarian reserve. The investigators aim is to measure ovarian reserve parameters in patients newly diagnosed with psoriasis and to compare them to healthy controls. Serum FSH,LH,E2,PRL and AMH will be measured on the 3rd day of the cycle.The serum hormone levels will be compared between women with psoriasis and women without psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Reproductive age group women: 18-40 years
* Women diagnosed with psoriasis (case group)
* Women without psoriasis (control group)

Exclusion Criteria:

* Women with PCOS (polycystic ovary syndrome)
* history of ovarian surgery
* Body mass index (BMI) over 30
* Women with other autoimmune diseases including Hashitomo thyroiditis
* Women with family history of premature ovarian insufficiency (POI)
* Women with infertility
* Psoriasis using systemic drugs including steroids and immunosuppressive therapy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Study Population: The study population will be reproductive age women diagnosed with psoriasis. The control population will be aged and BMI matched women without psoriasis.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
to compare serum AMH levels between the two groups | 1 day
  Serum AMH levels will be measured (using ELISA) and compared between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Berna Aslan Cetin, MD, Principal Investigator — Kanuni Sultan Suleyman Research and Training Hospital
Locations (1):
- Kanuni Sultan Suleyman Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: premature ovarian failure in patients with psoriasis — http://www.obgyn.net/asrm-2011/asrm-presentation-higher-risk-premature-ovarian-failure-and-early-menopause-cid